CLINICAL TRIAL: NCT04616261
Title: Trainability of the beta2-adrenergic System With Respect to Performance
Brief Title: Beta2-adrenergic System and Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: FOREX
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SET-HIGH (Experimental): High volume speed endurance training
  Interventions: Behavioral: Training; Drug: Formoterol; Drug: Placebo
- SET-LOW (Experimental): Low volume speed endurance training
  Interventions: Behavioral: Training; Drug: Formoterol; Drug: Placebo

INTERVENTIONS:
Behavioral: Training — 6 weeks of training
Drug: Formoterol — inhalation of 54 microg formoterol
Drug: Placebo — inhalation of placebo

SUMMARY:
This project aims to examine the trainability of the beta2-adrenergic system with respect to the individual performance response

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Trained individuals with a maximal oxygen uptake above 55 ml/min/kg
* Body mass index lower than 26

Exclusion Criteria:

* Allergy towards study drug
* Unacceptable side effects to the study drug
* Chronic disease deemed by the MD to interfere with the study
* Smoking
* Use of prescription medicine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2022-11-10 (Estimated); Study Completion 2022-11-10 (Estimated)

PRIMARY OUTCOMES:
Sprint performance | ½ hour after administration of formoterol or placebo
  Change in power output during maximal cycling in response to formoterol

SECONDARY OUTCOMES:
Cycling endurance performance | ½ hour after administration of formoterol or placebo
  Change in 4-min time trial performance in response to formoterol